CLINICAL TRIAL: NCT07288996
Title: Fractionated Spinal Anesthesia With Combined Isobaric and Hyperbaric Bupivacaine Toward Safer Anesthesia for Elderly Hip Fracture Patients: Randomized Controlled Study
Brief Title: Fractionated Spinal Anesthesia With Combined Isobaric and Hyperbaric Bupivacaine for Elderly Hip Fracture Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Salah Salem, Lecturer of anesthesia, Surgical intensive care and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR131034/10/25
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spinal Anesthesia in Elderly Patients
Keywords: Fractionated spinal anesthesia; hyperbaric bupivacaine; isobaric bupivacaine; hip fructure; elderly patients
MeSH Terms: interventions — DMAC2L protein, human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fractionated SA with isobaric and hyperbaric bupivacaine (Experimental): patients will receive fractionated SA in two doses first dose of hyperbaric bupivacaine with fentanyl followed after 90 seconds by the second dose of isobaric bupivacaine.
  Interventions: Procedure: Fractionated SA with isobaric and hyperbaric bupivacaine
- Fractionated SA with hyperbaric bupivacaine group (Active Comparator): patients will receive fractionated SA in two doses of hyperbaric bupivacaine and fentanyl, two thirds of the dose will be given firstly followed by the last third after 90 seconds.
  Interventions: Procedure: Fractionated SA with hyperbaric bupivacaine
- Conventional SA group (Active Comparator): patients will receive the conventional SA bolus dose of hyperbaric bupivacaine and fentanyl.
  Interventions: Procedure: Conventional SA group

INTERVENTIONS:
Procedure: Fractionated SA with isobaric and hyperbaric bupivacaine — patients will receive fractionated SA in two doses first dose of hyperbaric bupivacaine with fentanyl followed after 90 seconds by the second dose of isobaric bupivacaine.
  Other Names: Arm 1
  Arms: Fractionated SA with isobaric and hyperbaric bupivacaine
Procedure: Fractionated SA with hyperbaric bupivacaine — patients will receive fractionated SA in two doses of hyperbaric bupivacaine and fentanyl, two thirds of the dose will be given firstly followed by the last third after 90 seconds.
  Other Names: Arm 2
  Arms: Fractionated SA with hyperbaric bupivacaine group
Procedure: Conventional SA group — patients will receive the conventional SA bolus dose of hyperbaric bupivacaine and fentanyl.
  Other Names: Arm 3
  Arms: Conventional SA group

SUMMARY:
This prospective randomized controlled study will be conducted to compare the effect of fractionated SA using isobaric and hyperbaric bupivacaine with fractionated SA using hyperbaric bupivacaine and the conventional SA on hemodynamic instability in orthogeriatric patients undergoing hip fracture surgeries.

DETAILED DESCRIPTION:
Hip fractures are one of the most common reasons for elderly patients to present to the emergency department and require urgent surgery. Despite the debate regarding the preferred type of anesthesia in the elderly population, spinal anesthesia has shown the advantage of the simplicity of the technique, the better analgesic profile, the lower incidence of thromboembolic events and lower hospital stay. Hemodynamic stability should be considered as a primary intraoperative target. In pursuit of optimizing spinal anesthesia, this study proposed that fractionated SA by sequential administration of low doses of isobaric and hyperbaric bupivacaine can minimize hemodynamic instability while leveraging the advantages of both solutions when compared with fractionated SA using hyperbaric bupivacaine or the conventional SA technique.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients of both gender aged 65 years or more with American Society of Anesthesiologists (ASA) Physical Status I-III, who were scheduled for hip fracture surgeries under Spinal anesthesia

Exclusion criteria:

* Patients declined to participate in the trial.
* Patients on anticoagulation therapy.
* Patients planned for general anesthesia.
* Patients with atrial fibrillation.
* Allergies or hypersensitivity to local anesthetic drugs.
* Spinal cord deformities.
* Infection that contraindicate SA.
* Preoperative motor and sensory deficits

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | MAP will be measured intraoperatively before spinal anesthesia (SA), immediately after administering SA and subsequently at regular intervals 5, 10, 20, 30, 60, 75, 90 minutes, and then every 30 minutes till the end of surgery.
  Intraoperative hypotension is defined as the drop of systolic blood pressure (SBP) by 25% of the basal reading or the drop of MAP below 65 mmHg.

SECONDARY OUTCOMES:
Incidence of bradycardia. | HR will be measured intraoperatively before spinal anesthesia (SA), immediately after administering SA and subsequently at regular intervals 5, 10, 20, 30, 60, 75, 90 minutes, and then every 30 minutes till the end of surgery.
  Bradycardia is defined as sustained HR less than 60 beat/ minute
Vasopressor requirements. | intraoperatively after spinal anesthesia till the end of surgical intervention
  total dose of vasopressors required intraoperatively
Postoperative pain score | immediately post operatively then every 30 minutes up to 2 hour
  Visual analogue scale (VAS) is typically a 10-cm horizontal line labeled:
  * 0 = No pain
  * 10 = Worst imaginable pain
  A patient marks a point along the line to indicate their level of pain. The score is then measured in centimeters or millimeters to quantify pain intensity.
Time to first rescue analgesia | post operative .. time interval from the end of surgery until need of rescue analgesia
  time interval from the end of surgery until need of rescue analgesia

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available upon a reasonable request from the corresponding author after the end of the study for 1 year
Access Criteria: The data will be available upon a reasonable request from the corresponding author

REFERENCES:
- [Result] James LA, Levin MA, Lin HM, Deiner SG. Association of Preoperative Frailty With Intraoperative Hemodynamic Instability and Postoperative Mortality. Anesth Analg. 2019 Jun;128(6):1279-1285. doi: 10.1213/ANE.0000000000004085. PMID 31094800
- [Result] Meyhoff CS, Hesselbjerg L, Koscielniak-Nielsen Z, Rasmussen LS. Biphasic cardiac output changes during onset of spinal anaesthesia in elderly patients. Eur J Anaesthesiol. 2007 Sep;24(9):770-5. doi: 10.1017/S0265021507000427. Epub 2007 Apr 27. PMID 17462120
- [Result] Messina A, Frassanito L, Colombo D, Vergari A, Draisci G, Della Corte F, Antonelli M. Hemodynamic changes associated with spinal and general anesthesia for hip fracture surgery in severe ASA III elderly population: a pilot trial. Minerva Anestesiol. 2013 Sep;79(9):1021-9. Epub 2013 May 2. PMID 23635998
- [Result] Alrefaey AK, Bakrey SA. Sequential Intrathecal Injection of Hyperbaric and Isobaric Bupivacaine in Orthogeriatric Lower Limb Surgery, a Prospective Randomized Study. Asian J Anesthesiol. 2022 Jun 1;60(2). doi: 10.6859/aja.202206_60(2).0004. Epub 2022 May 4. PMID 35607733
- [Result] Niu Z, Xu X, Chu H, Yin J. Anesthetic management of hip fracture in geriatric patient with respiratory and heart failure using pericapsular nerve group block: A case report. Medicine (Baltimore). 2022 Jun 3;101(22):e29478. doi: 10.1097/MD.0000000000029478. PMID 35665737
- [Result] Carpintero P, Caeiro JR, Carpintero R, Morales A, Silva S, Mesa M. Complications of hip fractures: A review. World J Orthop. 2014 Sep 18;5(4):402-11. doi: 10.5312/wjo.v5.i4.402. eCollection 2014 Sep 18. PMID 25232517